CLINICAL TRIAL: NCT05317663
Title: Developing and Testing Waterpipe-specific Health Warning Labels Targeting Young People in Florida
Brief Title: Developing and Testing Waterpipe-specific Health Warning Labels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 20B16
Record Dates: First submitted 2022-02-28; First posted 2022-04-08 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Waterpipe Smoking; Health Warning Label; Harm Perception; Puffing Behaviour; Quitting Smoking; Health Risk Behaviors
Keywords: waterpipe; Health warning label; Young people
MeSH Terms: conditions — Water Pipe Smoking; Smoking Cessation; Health Risk Behaviors

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a 2x2x2x4 within-subject (2: HWL vs no-HWL x 2: pre- vs post- smoking) and between-subject (2: beginner vs established smokers x 4: HWLs) experimental study. Participant in each group (beginner, established smoker) will be randomly assigned to one of the 4 HWLs conditions, and undergo 2 WP smoking sessions that differ by HWL on the WP device (HWL vs. no-HWL), with pre-/post-smoking assessment of harm perception, intention to quit, puffing behavior, satisfaction, urge to smoke, and toxicant exposure. The investigators will use Latin Square crossover design balanced for carry-over effect (random order of 4 HWL condition), and to ensure equal distribution of study participants across gender.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waterpipe with Health Warning Label (HWL) (Experimental): All participants will complete a lab visit where they will smoke waterpipe with HWL for up to 45 minutes.
  Interventions: Behavioral: Test Health Warning Label (HWL)
- Absence of Waterpipe without Health Warning Label (HWL) (Experimental): All participants will complete a lab visit where they will smoke waterpipe without HWL for up to 45 minutes.
  Interventions: Behavioral: Test without Health Warning Label (no-HWL)

INTERVENTIONS:
Behavioral: Test Health Warning Label (HWL) — Effect of Health Warning Label (HWL)
  Arms: Waterpipe with Health Warning Label (HWL)
Behavioral: Test without Health Warning Label (no-HWL) — Effect of no Health Warning Label (no-HWL)
  Arms: Absence of Waterpipe without Health Warning Label (HWL)

SUMMARY:
Waterpipe (WP) smoking has become one of the leading tobacco use methods among youth in Florida. The impact of this dramatic rise is amplified by the mounting evidence of WP addictive and harmful nature, as well as the lag of policy response to it. Evidence suggests WP use leads to nicotine addiction, and increases the risk of lung cancer, heart and respiratory disease and exposure to secondhand smoke. The spread of WP use among youth has been fueled by a misperception of reduced-harm compared to cigarettes. Health Warning Labels (HWLs) represent one of the most successful tobacco control strategies to communicate smoking- related risks, and studies have consistently shown that HWLs are associated with a decrease in smoking rates and smoking-related morbidity and mortality. Therefore, communicating WP risks to young people through HWLs has been identified as a priority by major health bodies in the US including the FDA.

Using the Delphi method among international tobacco control experts, our team has developed a set of 12 WP HWLs corresponding to 4 health themes; health risks/addiction, harm to others, WP-specific harm, WP harm compared to cigarettes. Building on this work, and using a mixed- method approach incorporating qualitative and quantitative research, the investigators propose to:

Aim 1: Adapt the 12 HWLs to young WP smokers in Florida using exploratory focus groups.

Aim 2: Test in a clinical lab experiment the performance of the top 4 HWLs on the WP device compared to no-HWL/control on harm perception, intention to quit, and toxicant exposure (Carbon monoxide (CO), nicotine, oxidative stress).

Aim 3: Use the knowledge obtained to advocate for the adoption of WP-HWLs policies and disseminate information about WP harmful effects to young people in Florida and nationally.

Communicating WP risks through HWLs promises to reduce WP use and WP-related morbidly and mortality among young adults in Florida. This pioneering work will inform the FDA and public health advocates on the potential of WP-HWLs policies and provide a model for other states to respond to the WP epidemic.

DETAILED DESCRIPTION:
Our Team developed 12 pictorial Health Warning Labels (HWLs) for the waterpipe (WP) corresponding to 4 themes; health risks/addiction, harm to others, specific harm, and harm compared to cigarettes. The investigators will build on this work to advance HWLs policies and disseminate knowledge about WP harmful effects to young people in Florida and nationally through the following specific aims:

1. Adapt the HWLs to young adults in Florida using focus groups. The investigators will conduct mixed- gender focus groups combined with brief survey with regular WP smokers (6-8 groups; n ≈ 65; age 18-29 yrs) to 1- adapt the 12 HWLs to our target population, 2- explore their optimal placement and size, and 3- select the top 4 HWLs for testing (Aim 2).
2. Test the top 4 HWLs in a clinical lab experiment. Using the top 4 HWLs on the device, the investigators will recruit 2 groups of WP smokers (n= 248; age 18-29 yrs) based on their use frequency (beginners, established) for a within- (HWL vs no-HWL; pre- vs post- smoking) and between-subject (beginner vs. established; 4 HWLs) experiment. Participants will be randomly assigned to one of the 4 HWLs conditions and undergo 2 smoking sessions that differ by HWL (HWL vs. no-HWL), with pre-post smoking assessment of harm perception, intention to quit, and toxicant exposure. Participants will receive a follow-up phone call 3- month after exposure to assess longer-term changes in quit attitude and behavior. The investigators hypothesize that applying pictorial HWLs to the WP device will; 1- significantly increase harm perception and intention to quit, and reduce puffing behavior, satisfaction, and exposure to toxicants compared to no-HWL; 2- this effect will be more pronounced in beginner than established smokers.
3. Disseminate knowledge. The investigators will partner with Tobacco-Free Workgroup, and Truth Initiative to advocate for the adoption of HWLs policies and disseminate knowledge about WP harmful effects to young people in Florida and nationally.

Impact: Communicating WP risks through HWLs promises to reduce WP use and WP-related morbidly and mortality among young adults in the US.

ELIGIBILITY:
Inclusion Criteria:

* Age of 21-35 years.
* Beginners WP smokers (defined as started WP smoking in the past 6 months, but smoke WP less than weekly); or established WP smokers (defined as smoked at least once a week in the past 6 months).
* Generally healthy individuals (determined by physical examination).
* Is willing to provide informed consent.
* Is willing to attend the lab as required by the study protocol.
* Have abstained from WP for 12 hours prior to each lab session.

Exclusion Criteria:

* Women who are breast-feeding or test positive for pregnancy (by urinalysis at screening).
* Individuals with self-reported history of chronic disease or psychiatric conditions.
* Individuals with history of or active cardiovascular disease, low or high blood pressure, seizures, and regular use of prescription medications (other than vitamins or birth control).
* Report tobacco product use regularly (> 5 times/month in the past year).

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Intention and motivation to quit | pre-/post-smoking and at 3-month assessment. Each session is approximately 45 minutes ad lib use period.
  Intention and motivation to quit will be measured by using 3 items; "Does the participant intend to reduce WP smoking?"; "Does the participant intend to quit WP smoking?", and "How motivated is the participant to quit WP smoking in the next month?" The scale will be scored on a 5-point scale ranging from 1 (not at all), to 5 (very much).

SECONDARY OUTCOMES:
Harm perception | pre-/post-smoking and at 3-month assessment. Each session is approximately 45 minutes ad lib use period.
  Harm perception will be measured by using 1 item "To what extent does the participant think about the serious health effects of WP smoking?". This scale will assess WP harm perception and measure perceptions of WP relative risk compared to cigarettes. The scale will be scored on a 7-point scale ranging from 1 (not at all harmful), to 7 (extremely harmful).
Exhaled Breath Condensate (EBC) | It will be collected pre-post smoking session. Each session is approximately 45 minutes ad lib use period.
  To test for markers of oxidative stress and DNA damage. The investigators will test for 6 biomarkers (8-oxo-7,8-dihydro-2'-deoxyguanosine, 8-oxoguanosine, 8-isoprostane, formaldehyde, acetaldehyde and malondialdehyde). Samples will be collected during 15 min of tidal breathing through a single-use disposable Respiratory Tube Tympanic Membrane collector (Respiratory Research, Inc., Charlottesville, Va., USA). After sample collection, a plunger will be used to pool the condensed material within the tube into a single sample (about 1.0-2 ml). EBC samples will be divided in aliquots and stored at -80°C. EBC samples will be analyzed by our Forensic Chemistry Lab at Florida International University using Online Solid-Phase Extraction and Liquid Chromatography Triple Quadrupole Mass Spectrometry and Gas Chromatography Mass Spectrometry.
Social interaction | at 3-month assessment
  Social interaction will be measured by using 1 item "Since the participant started the study, how many times did the participant have a conversations with the family/friends about the HWLs?"
Change in WP smoking | at 3-month assessment
  Change in WP smoking will be measured by using 3 items; "Since the participant started the study, 1- did the participant stop smoking for 1 day or longer because the participant was trying to quit WP smoking?, 2- did the participant avoid smoking WP because the participant was thinking about the HWLs?, and 3- did the participant stop WP smoking completely because of the HWLs?"
Toxicant exposure: expired carbon monoxide | initially at the beginning of the smoking session (abstinence verification), and within 10 minutes after the WP smoking session
  expired carbon monoxide will be measured via expired carbon monoxide monitor.
Puff topography | continuously during smoking. Puffing behavior is continuously measured during each WP smoking session (an approximately 45 minutes ad lib use period)
  Measurement of puffing behavior.
Hear rate | continuously during smoking. Each session is approximately 45 minutes ad lib use period.
  Change in heart rate, measured in beats per minute.
Blood pressure | continuously during smoking. Each session is approximately 45 minutes ad lib use period.
  Change in blood pressure, measured in mm/hg.
Duke Sensory Questionnaire (DSQ) | DSQ will be measured only after smoking. The session is approximately 45 minutes ad lib use period.
  This scale will assess participants sensory experience of the inhaled product. The scale has nine items. All items will be scored on a 7-point Likert scale anchored at the extremes (1= not at all; 7=extremely).
The Cigarette/WP Evaluation Scale (WES) | WES will be measured only after smoking. The session is approximately 45 minutes ad lib use period.
  This scale assesses participants' perception of WP smoking. The scale has 11 items. All items will be scored on a 7-point Likert scale anchored at the extremes (1= not at all; 7=extremely).
Minnesota Nicotine Withdrawal Scale | During participants' 1st and 2nd visit. Questionnaire will be administered 2 times in each smoking session: before and after an approximately 45-min ad lib use period.
  This scale is used to assess the extent to which product use reduces tobacco abstinence symptoms, and consists of 11 items scored 0 - 100. These items are presented as Visual Analog Scale with item (measure) centered above a horizontal line anchored on the left with not at all and on the right with extremely.
Questionnaire of Smoking Urges | During participants' 1st and 2nd visit. Questionnaire will be administered 2 times in each smoking session: before and after an approximately 45-min ad lib use period
  This scale is used to assess the extent to which product use reduces tobacco abstinence symptoms, and consists of 10 items that are scored 0 - 7. Rated on a 7-point Likert scale ranging from 0 (strongly disagree) to 6 (strongly agree).
Lung function tests (LFTs) | During participants' 2 study visits. Lung function tests will be measured 2 times in each hookah smoking session: before and after an approximately 45 minutes ad lib use period
  LFTs (i.e., lung volume testing, airway resistance, specific airway conductance) will be measured before and immediately after hookah smoking. According to 2019 American Thoracic Society and European Respiratory Society recommendation simple spirometry (e.g., % predicted value pred (FVC), FEV1 % pred FEV1/FVC, % pred); forced expiratory flow (FEF) and peak expiratory flow rate or (PEFR) will be performed. Diffusing capacity for carbon monoxide (DLCO) will be determined using a rapidly resolving gas analyzer (RGA) and the single-breath technique. Note: This outcome is not involved in multiple assessments since all the values will appear on the spirometry at the same time.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/63/NCT05317663/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/63/NCT05317663/ICF_001.pdf